CLINICAL TRIAL: NCT00896376
Title: Prospective Multicenter Study of Genetic Factors Predictive of the Pharmacodynamics of Trastuzumab in Patients With Metastatic Breast Cancer
Brief Title: Trastuzumab in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000626782; CALACASS-2005/35; CALACASS-PHRC 2005 Herceptine; INCA-RECF0618
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (1):
- trastuzumab (Experimental)
  Interventions: Biological: trastuzumab; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: trastuzumab
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This clinical trial is studying the side effects of trastuzumab in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the predictive value of genetic factors on the toxicity and efficacy of a trastuzumab-based therapy in women with metastatic breast cancer.

Secondary

* To analyze tumor factors potentially related to the efficacy of trastuzumab (i.e., expression of proteins involved in cell proliferation and survival).

OUTLINE: This is a multicenter study.

Patients receive standard treatment with trastuzumab. Blood is collected periodically for pharmacogenetic analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic disease, defined by the existence of a secondary tumor localization radiologically (i.e., by radiography, CT scan, MRI scan, or ultrasound) or scintigraphically confrimed
* Evaluable disease
* Beginning first-line metastatic treatment with trastuzumab (Herceptin®) with or without chemotherapy
* Primary tumor must overexpress HER2 (IHC 3+ OR IHC 2+ and FISH+ OR FISH+)
* Hormone receptor status not specified
* No brain metastasis

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Life expectancy > 3 months
* Able to undergo cardiotoxicity evaluation every 4 months by measuring LVEF via an isotopic method or ultrasound with systematic registration
* No chronic uncontrolled disease
* No heart failure
* No respiratory failure or hypoxemia
* No history of another primary cancer except for basal cell carcinoma of the skin
* No severe uncontrolled infection
* No psychological incapacity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-12; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Toxicity, including cardiotoxicity and immuno-allergic reactions | 1 year
Clinical response as assessed by RECIST criteria | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Ferrero, MD, Study Chair — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France